CLINICAL TRIAL: NCT04229459
Title: A Phase II Study of the Addition of Nivolumab and Cetuximab to Chemoradiation in Locally Advanced Esophageal Squamous Cell Carcinoma (ESqCC).
Brief Title: Trial of Nivolumab and Cetuximab After Chemoradiation in Esophageal Squamous Cell Carcinoma Patients.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Baruch Brenner (Other)
Collaborators: Bristol-Myers Squibb (Industry); Merck Serono International SA (Industry)
Responsible Party: Sponsor-Investigator, Baruch Brenner, Director of the Oncology Division and the Davidoff Cancer Center, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-76W / MS062202_0103
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Cancer; Esophageal Squamous Cell Carcinoma; Cetuximab; Nivolumab
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Esophageal Neoplasms | interventions — Cisplatin; Fluorouracil; Radiotherapy; Cetuximab; Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Treatment (Experimental): All subjects will receive induction chemotherapy and chemoradiation combined with cetuximab followed by nivolumab and cetuximab as neoadjuvant treatment
  Interventions: Drug: Cisplatin; Drug: 5-FU; Radiation: Radiation therapy; Drug: Cetuximab; Drug: Nivolumab

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 100mg/m2 IV on day 1 of induction chemotherapy, 75mg/m2 IV on day 1 and 29 of chemoradiation
Drug: 5-FU — 5-FU 1000mg/m2/d IV on days 1-5 of induction chemotherapy, 1000mg/m2/d IV on days 1-4 and days 29-32 of chemoradiation
Radiation: Radiation therapy — 1.8 Gy/fraction, 5 days a week for a total of 28 days
Drug: Cetuximab — Cetuximab 400mg/m2 IV on day 1 followed by 250mg/m2 IV weekly on induction chemotherapy, 250mg/m2 IV weekly on chemoradiation, 500mg/m2 IV on day 1 of each treatment cycle, every two weeks during immunotherapy
  Other Names: Erbitux
Drug: Nivolumab — Nivolumab 3mg/kg IV on day 1 of each treatment cycle, every two weeks during immunotherapy
  Other Names: Opdivo

SUMMARY:
This is a phase II, open label, two-centered study for evaluation of the addition of nivolumab and cetuximab after chemoradiation as a neoadjuvant treatment for locally advanced esophageal squamous cell carcinoma patients. Subjects must have received no prior treatment for esophageal cancer (chemotherapy, radiotherapy or surgery) and no prior treatment with checkpoint inhibitors.

Eligible subjects will receive induction chemotherapy with cetuximab for a period of 4 weeks, chemoradiation with cetuximab for a period of 6 weeks, 3 cycles of immunotherapy (nivolumab + cetuximab) for a period of 6 weeks, and will undergo surgery at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written IRB approved informed consent.
* Age > 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Subjects with histologically confirmed operable, primary (non-recurrent) locally advanced (T3NxM0, TxN1M0) middle (distal to the thoracic inlet) or distal (up to the gastroesophageal junction) ESqCC according to endoscopic ultrasound (EUS) and PET-CT.
* No prior systemic or radiation therapy for esophageal cancer.
* Presence of adequate contraception in fertile patients.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
* Women must not be breastfeeding.
* No previous (within the last 5 years) or concurrent malignancies, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix or basal cell carcinoma of the skin.

Exclusion Criteria:

* Cervical esophageal tumors or tumors < 5 cm from the cricopharyngeal cartilage.
* Gastric cancers with minor involvement of the GEJ or distal esophagus, or an esophageal tumor extending beyond 2 cm into the stomach.
* Prior chest or upper abdomen radiotherapy, prior systemic chemotherapy within the past 5 years or prior esophageal or gastric surgery.
* Patients with evidence of metastatic disease.
* Biopsy proven tumor invasion of the tracheobronchial tree or presence of tracheo-esophageal (TE) fistula or recurrent laryngeal nerve or phrenic nerve paralysis.
* New York Heart Association Class III or IV heart disease. Angina or myocardial infarction within the last 12 months, history of significant ventricular arrhythmia requiring medication with antiarrhythmics, or a history of a clinically significant conduction system abnormality.
* Clinically significant hearing loss.
* Patients with a history of seizure disorder who are receiving phenytoin, phenobarbital, or other antiepileptic medication.
* Any positive test for hepatitis B virus or hepatitis C virus indicating active infection.
* Ongoing immunosuppressive therapy.
* Active autoimmune disease. [Subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll].
* Prior organ transplant.
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Known history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2027-04-04 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) rate | Time from start of neoadjuvant treatment until surgical resection, assessed up to 24 months
  pCR is defined when no tumor is found on pathology review of the surgical specimen (TRG -0)
Modified pathological complete response | Time from start of neoadjuvant treatment until surgical resection in operated patients (pCR) and long-term (≥12 months) clinical complete response (cCR) in unoperated patients, assessed up to 24 months.
  We defined a novel primary endpoint, combining pathological complete response (pCR) rate among operated patients and long-term (≥12 months) clinical complete response (cCR) rate for those electing watchful waiting, into a composite endpoint of modified pCR (mpCR) rate.
Progression Free Survival (PFS) | The time interval from the first day of treatment to the first event of loco-regional failure, metastatic recurrence or death from any cause, assessed up to 66 months
  PFS will be censored in patients without loco-regional failure, metastatic recurrence or death, at the last date known to be alive or at the start of a new anti-cancer treatment, whatever occurs first. PFS rate will be estimated using the Kaplan-Meier method
Incidence of Treatment-Emergent Adverse Events (Safety) | Time from screening until the end of study drug administration, assessed up to 24 months
  Treatment-emergent AEs will be graded according to NCI CTCAE v5.0, vital signs and clinical laboratory

SECONDARY OUTCOMES:
Overall survival (OS) | The time interval between the first day of treatment and the date of death from any cause, assessed up to 66 months
  Patients who are still alive when last traced will be censored at the date of last follow-up. OS rate will be estimated using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Baruch Brenner, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel